CLINICAL TRIAL: NCT05561777
Title: Implementation of Penicillin Allergy Risk Stratification and Delabeling of Low-Risk Patients: Provider-Targeted Clinical Decision Support Versus Pharmacist-Led Approach
Brief Title: Penicillin Allergy Risk-Stratification and Delabeling of Low-Risk Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: screening challenges that prevented the intervention from being implemented
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, James Antoon, Assistant Professor of Pediatrics, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 220060
Record Dates: First submitted 2022-09-26; First posted 2022-09-30 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Antibiotic Allergy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pharmacist-led Evaluation (No Intervention): Patients randomized to the pharmacist-led arm will appear in the pharmacy-penicillin electronic health care dashboard. A pharmacist may, at their discretion and in consultation with the primary care team, perform an allergy risk-stratification and oral challenge in low-risk patients using local standard of care protocol
- Provider-targeted Clinical Decision Support Tool (Experimental): This intervention will provide access to a best-practices alert (BPA) containing the patient's risk-stratification status and a link to the local standard of care protocol, oral amoxicillin challenge order set and written consent form (same resources as used in pharmacist -led electronic health record dashboard). If the provider opts to perform the oral challenge and it is successfully passed, a second BPA will prompt them to update the allergy status in the medical record.
  Interventions: Other: Physician-targeted CDS tool for PCN allergy delabeling

INTERVENTIONS:
Other: Physician-targeted CDS tool for PCN allergy delabeling — This intervention will provide access to a best-practices alert (BPA) containing the patient's risk-stratification status and a link to the local standard of care protocol, oral amoxicillin challenge order set and written consent form (same resources as used in pharmacist -led electronic health record dashboard). If the provider opts to perform the oral challenge and it is successfully passed, a second BPA will prompt them to update the allergy status in the medical record.
  Arms: Provider-targeted Clinical Decision Support Tool

SUMMARY:
Children are often reported to have antibiotics allergies, with approximately 10% of the US population labeled as allergic to an antibiotic, however, recent studies have demonstrated that the majority of symptoms reported as an allergy by parents are often non-IgE-mediated adverse reactions or symptoms of a viral illness (e.g. rash, vomiting, diarrhea). Additionally, over 90% of patients with reported penicillin allergy have negative skin testing results. Several studies in children have found that an allergy questionnaire can accurately identify those who are at low risk for severe antibiotic allergy and the allergy label can be safely removed. Appropriately delabeling antibiotic allergies has been shown to improve patient care through changing prescribing behavior and lowering health care costs.

In this study, the investigators will perform a randomized trial comparing a provider-targeted clinical decision support tool to a pharmacist-led approach. The physician-targeted CDS tool will inform providers of their patient's allergy risk stratification result, protocol, electronic health record order and documentation support. The pharmacist-led approach consists of electronic health record dashboard that includes identical information to the provider arm. The primary outcome will be the frequency of penicillin allergy encounters with an allergy label removed at the time of discharge. Secondary outcomes will include the percentage of encounter with a penicillin allergy label in the electronic medical record 3 months after discharge, hospital length of stay and antibiotic utilization.

ELIGIBILITY:
Inclusion Criteria:

Pediatric Hospital Medicine service Existing penicillin allergy label in the EHR Screened as low-risk for true PCN allergy (based on usual-care nursing intake questions at time of admission)

Exclusion Criteria:

None, provider may opt out of CDS tool at any time

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Allergy Delabeling Performed | Within 1 day of discharge for each encounter
  Percentage of enrolled encounters (intervention arm) in which providers perform allergy delabeling

SECONDARY OUTCOMES:
Allergy Label Adjustments in EHR | 3 months after discharge for each encounter
  Percentage of enrolled encounters with an oral challenge in which allergy label has been removed from patients' medical records.

CONTACTS AND LOCATIONS:
Overall Officials: James Antoon, MD, PhD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Monroe Carell Jr Children's Hospital at Vanderbilt, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No